CLINICAL TRIAL: NCT04419883
Title: Provider Satisfaction of a New, Flexible Extended-Length Pharyngeal Airway to Relieve Upper Airway Obstructive During Deep Sedation: A Pilot Study
Brief Title: A New Flexible Extended-Length Pharyngeal Airway for Deep Sedation
Status: Completed | Type: Observational
Sponsor: McMurray Medical Group, LLC (Industry)
Responsible Party: Principal Investigator, Roxanne R McMurray, VP of Clinical Management, McMurray Medical Group, LLC
Other Study IDs: MEA-001-01
Record Dates: First submitted 2020-05-29; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Upper Airway Obstruction
Keywords: Upper airway obstruction; Airway management tools; Airway complications; Deep sedation; Deep monitored anaesthesia care (MAC)
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Anesthesia Providers: Anesthesia providers from 15 different health care facilities in the United States.
  Interventions: Device: McMurray Enhanced Airway

INTERVENTIONS:
Device: McMurray Enhanced Airway — Provider Satisfaction of a New, Flexible Extended-Length Pharyngeal Airway to Relieve Upper Airway Obstructive During Deep Sedation: A Pilot Study
  Other Names: MEA

SUMMARY:
The purpose of this prospective pilot provider adoption study was to evaluate user experience a new airway device in adult patients with airway obstruction under deep sedation. Fifteen hospital systems served as testing sites. Fifty-four anaesthetist providers reported their experience with the airway device in 84 cases across two phases of surveying.

DETAILED DESCRIPTION:
This multi-center proof-of-concept, descriptive, prospective, and observational study was approved by a universal Institutional Review Board (IRB) for Human Subjects Research in March 2019. Anaesthesia providers who volunteered to trial this new airway device were recruited to complete a survey tool to assess provider satisfaction of a commercially-available upper airway device (McMurray Enhanced Airway (MEA); McMurray Medical, Minneapolis, MN).

The MEA is a novel upper airway device with numerous enhanced features relative to currently available airway management products (Figure 1). The MEA has longer flexible tubing allowing for displacement of pharyngeal tissue that oral airways are unable to reach, and avoiding the need for chin lift/jaw thrust maneuvers [16]. The smaller diameter helps reduce stimulation and gagging and permits placement alongside an endoscopy bite block. The softer material, similar to that of a nasal airway, allows for ease of insertion and reduces potential oral injury associated with hard plastic oral airways [16]. An elongated cushioned bite block is designed to prevent proximal airway collapse, allow flexibility of molar placement, and decrease the risk of dental damage [16]. An optional connector can be connected to an anesthesia circuit or manual resuscitator, facilitating intraoral ventilation and aiding in situations such as difficult mask ventilation or when oxygen diffusion in the surgical field may present fire risk [16]. Furthermore, the MEA was designed to reduce need for manual stationary maneuvers by providers such as chin lift or jaw thrust, thereby preventing potential provider-patient exposure of airborne droplets and increased staffing.

Providers received device instructions for use (IFU) by training video and printed material to understand how to use and size the MEA. After using the MEA trial device in clinical practice, anaesthesia providers participated in completing the Use Survey Tool based on cases meeting the following criteria: inclusion criteria included adult patients (age >18) experiencing an obstructive airway under deep sedation; exclusion criteria included determining that the device size was inappropriate-too big or small-for the patient, since placing an improper size could be detrimental for the patient.

The initial survey(Phase 1) was developed to evaluate current product usage, general use conditions, deep sedation conditions, general anaesthesia conditions, device performance, and overall device satisfaction using binary responses with option for subjective free response. Based on Phase 1 responses and provider feedback, Phase 2 surveys were limited to questions with ordinal responses that assessed device use satisfaction during deep sedation procedures only. Surveys were distributed with the trial devices. As this was a pilot feasibility study for the new extended pharyngeal airway device, recruitment of provider subjects was based on interest of using a novel airway device to benefit airway management when providing deep sedation in situations where airway obstruction became problematic. Surveys were voluntarily completed by the anaesthesia provider following each use. One provider could complete multiple surveys to represent individual device performance and experience. Information related to patient, provider, and device placement frequency was not collected in order to expedite response rate to learn initial provider experience. Submitted surveys underwent response analysis by an independent statistician. Due to the nature of qualitative data, descriptive statistics were used to summarize study results. No objective measures of device clinical efficacy were collected.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Scheduled for surgery with sedation/MAC anesthesia
* Patients experiencing an obstructive airway needing an airway device placed

Exclusion Criteria:

• Inappropriate airway device size, too big or too small

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Anesthesia providers who volunteered to trial this new airway device were recruited to complete a survey tool to assess provider satisfaction of a commercially-available upper airway device (McMurray Enhanced Airway (MEA); McMurray Medical, Minneapolis, MN).
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the new, flexible extended-length pharyngeal airway ease of use | Survey was completed immediately after completion of surgery and airway use
  The question asked: With the curve end facing the hard palate, how easy was the MEA to place? Four response options on measurement tool to assess outcomes: Easy, Moderate, Difficult, Not Successful
Assess the new, flexible extended-length pharyngeal ability to relieve an upper airway obstruction | Survey was completed immediately after completion of surgery and airway use
  Two response options on measurement tool to assess outcomes: Yes and No
Assess if the new airway allowed a "hands off approach" when the patient was under deep sedation/MAC anesthesia | Survey was completed immediately after completion of surgery and airway use
  Three response options on measurement tool to assess outcomes: Yes, No, Not sure

SECONDARY OUTCOMES:
Provider satisfaction with the new, flexible extended-length pharyngeal airway. | Survey was completed immediately after completion of surgery and airway use
  Five response options on measurement tool to assess outcomes: Very Satisfied, Somewhat Satisfied, Satisfied, Dissatisfied, I did not use the MEA for deep MAC

CONTACTS AND LOCATIONS:
Overall Officials: Roxanne McMurray, DNP, Principal Investigator — McMurray Medical Group, LLC
Locations (1):
- Roxanne McMurray, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data was collected for this study